CLINICAL TRIAL: NCT02726984
Title: Assessment of Symptomatic and Asymptomatic Carotid Plaques Using Hybrid Imaging 18F-sodium Fluoride PET/MR
Brief Title: Carotid Plaque Assessment Using 18Fluorine (18F) -Sodium Fluoride Positron Emission Tomography (PET) /MR
Acronym: CARTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL15_0283; 2015-002327-26 (EudraCT Number)
Record Dates: First submitted 2015-12-15; First posted 2016-04-04 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Carotid Artery Plaque
Keywords: stroke; carotid plaque; 18F-sodium fluoride PET/MR
MeSH Terms: conditions — Carotid Stenosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- case (Experimental): Patients with carotid plaque ≥ 50% symptomatic (ischemic stroke on CT or MR) during the last 15 days
  Interventions: Drug: 18F-sodium fluoride PET/MR
- control (Experimental): Patients with asymptomatic carotid plaque ≥ 50%
  Interventions: Drug: 18F-sodium fluoride PET/MR

INTERVENTIONS:
Drug: 18F-sodium fluoride PET/MR — 18F-sodium fluoride PET/MR combining 3Tesla (3T) MR and PET producing 127 slices of 2 mm on an axial field of view of 26 cm. 18F-sodium fluoride (2 à 4 megabecquerel/kilogram (MBq/kg)) will be injected 60 min before.

SUMMARY:
Carotid plaque can lead to ischemic stroke. Treatment of asymptomatic carotid plaque, based on degree stenosis, is still controversial. Beyond the degree of stenosis, the composition of the plaque could reflect the vulnerability and the risk of ipsilateral ischemic stroke. Identification of new predictive factor of ipsilateral ischemic stroke in patients with carotid plaque could help to screen high risk patients and to guide the treatment. The aim of the study is to assess 18F-sodium fluoride uptake among carotid plaque in recently symptomatic and asymptomatic patients. Investigators conduct a pilot case-control study. Twelve patients (6 recently symptomatic and 6 asymptomatic) with carotid stenosis (≥50% NASCET) will have a 18F-sodium fluoride PET/MR. Standardized uptake value (SUV) and tissue-to-background ratio (TBR) will be measured among carotid plaques.

ELIGIBILITY:
Inclusion Criteria symptomatic patients:

* age>18
* Carotid plaque ≥ 50% symptomatic (ischemic stroke on CT or MR) during the last 15 days or asymptomatic
* ability to give informed consent
* affiliation to social security

Exclusion Criteria:

* Modified Rankin score ˃ 3
* Contraindication to MRI
* Renal failure (creatinine clearance by cockcroft ˂ 50 ml / min)
* Pregnancy / Breastfeeding
* Hypersensitivity to the active substance or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Measure of SUV (standardized uptake value) among carotid plaques ≥ 50% | during the last 15 days in symptomatic patients
Measure of TBR (tissue-to-background ratio) among carotid plaques ≥ 50% | at day 0 in asymptomatic patients
Measure of SUV (standardized uptake value) among carotid plaques ≥ 50% | at day 0 in asymptomatic patients
Measure of TBR (tissue-to-background ratio) among carotid plaques ≥ 50% | during the last 15 days in symptomatic patients

SECONDARY OUTCOMES:
Number of participants with image of lipid-rich necrotic core accounting for more than 50% of the surface of the plate on a 2D section. | during the last 15 days in symptomatic patients
  identification of images of intraplaque hemorrhage (defined as an hyperintense region within the plaque on a T1-weighted sequence), lipid-rich necrotic core (accounting for more than 50% of the surface of the plate on a 2D section), or thinning/rupture of the fibrous cap (identified on a T1-weighted sequence following intravenous gadolinium administration) in High Resolution MRI by two radiologists.
Number of participants with image of intraplaque hemorrhage defined as an hyperintense region within the plaque on T1-weighted sequence. | during the last 15 days in symptomatic patients
  identification of images of intraplaque hemorrhage (defined as an hyperintense region within the plaque on a T1-weighted sequence), lipid-rich necrotic core (accounting for more than 50% of the surface of the plate on a 2D section), or thinning/rupture of the fibrous cap (identified on a T1-weighted sequence following intravenous gadolinium administration) in High Resolution MRI by two radiologists.
Number of participants with image of thinning/rupture of the fibrous cap on a T1-weighted sequence following intravenous gadolinium administration. | during the last 15 days in symptomatic patients
  identification of images of intraplaque hemorrhage (defined as an hyperintense region within the plaque on a T1-weighted sequence), lipid-rich necrotic core (accounting for more than 50% of the surface of the plate on a 2D section), or thinning/rupture of the fibrous cap (identified on a T1-weighted sequence following intravenous gadolinium administration) in High Resolution MRI by two radiologists.
Number of participants with image of lipid-rich necrotic core accounting for more than 50% of the surface of the plate on a 2D section. | at day 0 in asymptomatic patients
  identification of images of intraplaque hemorrhage (defined as an hyperintense region within the plaque on a T1-weighted sequence), lipid-rich necrotic core (accounting for more than 50% of the surface of the plate on a 2D section), or thinning/rupture of the fibrous cap (identified on a T1-weighted sequence following intravenous gadolinium administration) in High Resolution MRI by two radiologists.
Number of participants with image of thinning/rupture of the fibrous cap on a T1-weighted sequence following intravenous gadolinium administration. | at day 0 in asymptomatic patients
  identification of images of intraplaque hemorrhage (defined as an hyperintense region within the plaque on a T1-weighted sequence), lipid-rich necrotic core (accounting for more than 50% of the surface of the plate on a 2D section), or thinning/rupture of the fibrous cap (identified on a T1-weighted sequence following intravenous gadolinium administration) in High Resolution MRI by two radiologists.
Number of participants with image of intraplaque hemorrhage defined as an hyperintense region within the plaque on T1-weighted sequence. | during the last 15 days in symptomatic patients
  Quantitative assessement of the wall shear stresses (WSS, measured in Pa) and oscillatory shear indexes (OSI, unitless) along the carotid wall in 3D. An accurate analysis of the hemodynamic environment will be performed using fluid dynamics mathematical models that allow the calculation of hemodynamic stress at the plate (or "wall shear stress" measured in Pascal) and temporal oscillation of the direction of this force (arbitrary units).
Quantitative assessement of the wall shear stresses (WSS, measured in Pa) along the carotid wall in 3D. | at day 0 in asymptomatic patients
  Quantitative assessement of the wall shear stresses (WSS, measured in Pa) along the carotid wall in 3D. An accurate analysis of the hemodynamic environment will be performed using fluid dynamics mathematical models that allow the calculation of hemodynamic stress at the plate (or "wall shear stress" measured in Pascal) and temporal oscillation of the direction of this force (arbitrary units).
Quantitative assessement of oscillatory shear indexes (OSI, unitless) along the carotid wall in 3D. | at day 0 in asymptomatic patients
  Quantitative assessement of oscillatory shear indexes (OSI, unitless) along the carotid wall in 3D. An accurate analysis of the hemodynamic environment will be performed using fluid dynamics mathematical models that allow the calculation of hemodynamic stress at the plate (or "wall shear stress" measured in Pascal) and temporal oscillation of the direction of this force (arbitrary units).
Number of participants with histological image of intraplaque hemorrhage, and/or lipid-rich necrotic core and /or thinning/rupture of the fibrous cap in surgical patients. | during the last 15 days in symptomatic patients
Measure of systemic markers of inflammation: Interleukine 1-Beta (IL1-beta), Tumor Necrosis Factor-alpha (TNF-alpha) | at Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Norbert NIGHOGHOSSIAN, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mechtouff L, Sigovan M, Douek P, Costes N, Le Bars D, Mansuy A, Haesebaert J, Bani-Sadr A, Tordo J, Feugier P, Millon A, Luong S, Si-Mohamed S, Collet-Benzaquen D, Canet-Soulas E, Bochaton T, Crola Da Silva C, Paccalet A, Magne D, Berthezene Y, Nighoghossian N. Simultaneous assessment of microcalcifications and morphological criteria of vulnerability in carotid artery plaque using hybrid 18F-NaF PET/MRI. J Nucl Cardiol. 2022 Jun;29(3):1064-1074. doi: 10.1007/s12350-020-02400-0. Epub 2020 Nov 3. PMID 33145738